CLINICAL TRIAL: NCT04538183
Title: Use Test: Dermowas Body Lotion pH 4 vs. pH 5.8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DK-01/2017
Record Dates: First submitted 2020-08-27; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Exploratory, Randomized, Double-blind (regarding the two test products), Intra-individual comparison
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The test areas were 5 x 5 cm squares on both inner (volar) forearms. The areas were randomized and double-blinded (regarding the two test products). For randomization, the permutated orthogonal Latin square method was used on condition that both test areas are always contralateral.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WO 5000 (Experimental): Body lotion pH 4 for topical application
  Interventions: Other: WO 5000
- WO 5001 (Experimental): Body lotion pH 5.8 for topical application
  Interventions: Other: WO 5001
- No product use (No Intervention): Untreated control area

INTERVENTIONS:
Other: WO 5000 — WO 5000
  Arms: WO 5000
Other: WO 5001 — WO 5001
  Arms: WO 5001

SUMMARY:
The objective of the study was to examine whether normalizing of the pH by acidification through topical treatment helps to strengthen the skin barrier, to induce epidermal differentiation and to reduce inflammation in healthy individuals.

DETAILED DESCRIPTION:
Previous studies have shown that an emollient adjusted to pH 4 has favorable effects to the skin of aged individuals. The objective of the study was to examine whether normalizing of the pH by acidification through topical treatment helps to strengthen the skin barrier, to induce epidermal differentiation and to reduce Inflammation. The effect of a cosmetic oil-in-water (O/W) emulsion adjusted to pH 4 in comparison to the same emulsion adjusted to pH 5.8 on the integrity of the skin barrier and the mechanical stability was examined in healthy volunteers from age 18 to 75 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers (75 % women and 25 % men)
* Aged 18 - 75 years
* Healthy skin
* Informed consent was given

Exclusion Criteria:

* Atopic diathesis, atopic dermatitis and other skin diseases with a disrupted skin barrier
* Dermatitis and other skin diseases in the test site
* Birthmarks, tattoos, scars and other abnormalities in the test site, which may influence the measurements
* Women: pregnancy and breastfeeding
* Known contact sensitization
* Severe systemic diseases
* Regular use of sauna and solarium
* Intensive UV exposure
* Topical use of drugs in the test site four weeks before and during the study
* Systemic administration of anti-inflammatory, immune-modulating and antibiotic drugs
* Previous participation in other studies within the last month before the study
* Alcohol and drug misuse
* Missing awareness and inability to follow the instructions of the study staff
* Other reasons which according to the study leader speak against the participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change of transepidermal water loss (TEWL) | Change from day 1 (before application) to day 30
  Tewameter TM300, Courage & Khazaka, Köln
Change of skin hydration | Change from day 1 (before application) to day 30
  Corneometer CM 825, Courage & Khazaka, Köln
Change of erythema | Change from Day 1 to day 30 + 2 hours (after tape-stripping), measured over 3 timepoints (Day 1, day 30 and day 30 +2 hours (after tape stripping)
  Visible score adapted from Frosch and Kligman: 0 = no redness, 0.5 = very slight redness, 1 = slight patchy or diffuse redness, 2 = moderate even redness, 3 = profound redness
Change of pH | Change from Baseline to day 31, measured over 5 time points (Day 1, day 30, day 30+3 hours, day 30+6 hours and day 31)
  pH-Meter 910, Courage & Khazaka, Köln
Tape-stripping | Day 31
  Number of the tape-strips until a threefold increase in TEWL compared to unstripped baseline value is reached. (D-Squame® (DSQ), CuDerm Corporation, Dallas)
Corneocyte size | Day 31
  After staining with Nile Red by immunofluorescence microscopy and digital imaging
Amount of the cytokine IL-1α | Day 31
  Determined by enzyme-linked immunosorbent assay (ELISA)
Amount of antimicrobial peptide hBD-2 | Day 31
  Determined by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Sören Merker, Dr., Study Chair — Dr. August Wolff GmbH & Co. KG Arzneimittel
Locations (1):
- Universitäts-Hautklinik Kiel, Kiel, Schleswig-Holstein, Germany